CLINICAL TRIAL: NCT03647787
Title: Changes of White Matter Integrity According to BDNF Genotype During Motor Recovery After Stroke
Brief Title: White Matter Integrity According to BDNF Genotype After Stroke
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-04-146
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2018-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — brain-derived neurotrophic factor (BDNF) genotype single nucleotide polymorphism (SNP): a methionine (Met) substitution for valine (Val) at codon 66 (Val66Met; rs6265)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — This study is a longitudinal observational study

SUMMARY:
The aim of this study was to investigate differential plastic changes of fractional anisotropy (FA) in the corticospinal tract (CST), the intrahemispheric corticocortical tract from the primary motor cortex to ventral premotor cortex (M1PMv) and the corpus callosum (CC) from 2 weeks to 3 months after stroke according to BDNF genotype.

DETAILED DESCRIPTION:
The aims of this study were to investigate plastic changes in the fractional anisotropy (FA) of three motor-related white matter fibers according to the BDNF genotype from 2 weeks to 3 months after stroke onset; one is a the majority of fibers from M1 to medullary oblongata (CST), another is the intrahemispheric connection from M1 to ventral premotor cortex (M1PMv), and the other is the interhemispheric connection between bilateral M1s (CC). There were also to investigate the relationships between motor impairment and tract-related FA of white matter tracts in each BDNF genotype

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with first-ever hemispheric ischemic infarction with damage to the supratentorial area confirmed by brain MRI within 2 weeks after stroke onset

Exclusion Criteria:

* any clinically significant or unstable medical disorder or neuropsychiatric comorbidity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke who were admitted to Samsung Medical Center and transferred to the Department of Physical and Rehabilitation Medicine
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy | 2 weeks to 3 months after stroke onset
  changes of fractional anisotropy (FA) in the corticospinal tract (CST)

SECONDARY OUTCOMES:
Fractional anisotropy | 2 weeks to 3 months after stroke onset
  changes of fractional anisotropy (FA) in the intrahemispheric corticocortical tract from the primary motor cortex to ventral premotor cortex (M1PMv)
Fractional anisotropy | 2 weeks to 3 months after stroke onset
  changes of fractional anisotropy (FA) in the corpus callosum (CC)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park E, Lee J, Chang WH, Lee A, Hummel FC, Kim YH. Differential Relationship between Microstructural Integrity in White Matter Tracts and Motor Recovery following Stroke Based on Brain-Derived Neurotrophic Factor Genotype. Neural Plast. 2020 Sep 22;2020:5742421. doi: 10.1155/2020/5742421. eCollection 2020. PMID 33029116